CLINICAL TRIAL: NCT04735354
Title: Sacubitril/Valsartan in Heart Failure With Reduced Ejection Fraction Patients: a Real World Study in India
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BIN01
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
Keywords: heart failure with reduced ejection fraction; HFrEF; India; sacubitril; valsartan; electronic medical records; EMRs; retrospective; RWE
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sacubitril/valsartan: Patients administered sacubitril/valsartan by prescription
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — There was no treatment allocation. Patients administered sacubitril/valsartan by prescription that started before inclusion of the patient into the study were enrolled.

SUMMARY:
This was a non-interventional, retrospective EMR analysis of longitudinal prescriptions in India for a period of 1.5 years. Demographic profile of patients with heart failure with reduced ejection fraction on sacubitril/valsartan was recorded.

DETAILED DESCRIPTION:
Index date was date of 1st prescription of sacubitril/valsartan. Dose titration of sacubitril/valsartan was assessed for a period of 6 months post index date.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with a diagnosis of HFrEF as mentioned in database or heart failure with a recording of LVEF <40% at or before the index date
* A prescription of sacubitril/valsartan

Exclusion Criteria:

* Diagnosis of HF specified as preserved/mid-range ejection fraction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years with a diagnosis of HFrEF as mentioned in database or heart failure with a recording of LVEF <40% at index date with a prescription of sacubitril/valsartan
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Age information | Index date
  Age information was reported
Gender information | Index date
  Gender information was reported
Number of participants by Geographic area | idex date
  Geographic area divided into 4 zones- North, South, East and West
Functional Class (New York Heart Association (NYHA) classification) | index date
  The New York Heart Association Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
Body Mass Index | Index date
  Median value body mass index was reported
Classification of Heart Failure by etiology | 1.5 years
  Coronary artery disease, valvular, rheumatic heart disease, others, unknown.
Change in ventricular function defined by Left Ventricular Ejection Fraction (LVEF) | Index date, 1.5 years
  An ejection fraction (EF) is the volumetric fraction (or portion of the total) of fluid ejected from a chamber with each contraction (or heartbeat).
Medical History | 1.5 years
  type 2 diabetes, chronic obstructive pulmonary disease (COPD), anemia, chronic renal disease, atrial fibrillation, stroke, hypertension, myocardial infarction
Number of participants with notable changes in laboratory parameters | Baseline, 1.5 years
  Safety measured by the notable post-baseline changes in laboratory parameters compared to baseline
Number of Hospitalizations | 1.5 years
  Hospitalizations due to cardiovascular and non-cardiovascular causes
Number of participants with concomitant medications | up to 6 months pre index date, Up to 6 months post index date
  Concomitant medications classified as-
  * Medications for HF: Diuretics, digitalis, beta-Blockers, ACEi, ARBs, MRA, ivabradine, SGLT2 inhibitors.
  * Medications for non-HF conditions: Anti-diabetic medications other than SGLT2 inhibitors (oral and injectable), statin, antiplatelet therapy, oral anti-coagulants.
Number of patients with other treatments for heart failure | 1.5 years
  Other treatments for heart failure like implantable cardioverter-defibrillator (ICD), and cardiac resynchronization therapy (CRT).

SECONDARY OUTCOMES:
Persistence to sacubitril/valsartan | Up to 12 months post index date
  Defined as time duration from initiation to discontinuation of therapy.
Proportion of patient discontinuing sacubitril/valsartan | month 2, month 4, month 6, month 8 and month 12
  Reported as frequency (n) and percentage (%).
Maximum individual dose reached | 6 months post index date
  Median value of maximum individual dose reached will be reported
Time to first dose up-titration | 6 months post index date
  Median time to first dose up-titration
Time to target dose | 6 months post index date
  Median time to target dose
Individual dose | 6 months post index date
  The proportion of patients with a starting dose of 50 mg, 100 mg, 200 mg
Titration patterns | 1.5 years
  Listings for all titration patterns which evaluated longitudinally at the patient level as follows:
  * Up-titration' corresponds to all patients who experience an initial increase in sacubitril/valsartan dose post-index,
  * 'Stable up-titration' corresponds to up-titrated patients who experience no subsequent decrease in sacubitril/valsartan dose
  * 'Down-titration' corresponds to all patients who experience an initial dose decrease in sacubitril/valsartan dose post-index, and
  * 'Stable down-titration' corresponds to the proportion of down-titrated patients who experience no subsequent up-titration.
Proportion of patients being titrated to 100mg from 50mg | 1.5 years
  Proportion of patients being titrated to 100mg from 50mg
Proportion of patients being titrated to 200mg from 100mg | 1.5 years
  Proportion of patients being titrated to 200mg from 100mg

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Mumbai, India

IPD SHARING:
Plan to Share IPD: No